CLINICAL TRIAL: NCT02212418
Title: Effect of an Abdominal Hypopressive Technique Program on Pelvic Floor Muscles and Urinary Incontinence in Women: A Randomized Cross-over Trial
Brief Title: Effect of an Abdominal Hypopressive Technique Program on Pelvic Floor Muscles and Urinary Incontinence in Women
Acronym: UVa_1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rafael J. Curbelo (Other)
Responsible Party: Sponsor-Investigator, Rafael J. Curbelo, PhD, University of Valladolid
Organization: University of Valladolid (Other)
Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: UValladolid_1
Record Dates: First submitted 2014-08-02; First posted 2014-08-08 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: Mild Pelvic Floor Dysfunction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Abdominal hypopressive technique (Experimental)
  Interventions: Other: Abdominal hypopressive technique

INTERVENTIONS:
Other: Abdominal hypopressive technique — postural technique based on self-elongating, body axis anteriorization, shoulders extension, and maintenance of an expiratory apnea as long as possible

SUMMARY:
Abdominal hypopressive technique (AHT) is a therapy created for the treatment of the pelvic floor dysfunctions in the postpartum. In the last years it has been extended out of such medical context but there is a lack of scientific evidence, and the endurability of the effects of this technique are unknown. The investigator´s aim was to evaluate the effect of a 12 weeks AHT program on 1) the tone of the pelvic floor muscles and 2) on urinary incontinence, in women out of the postpartum phase. In addition the investigators looked for the endurability of its effect.

Methods: The investigators performed a cross-over blinded intervention study of 4 month duration, in which women, stratified by age, were randomly assigned to a sequence of AHT-no AHT or no AHT-AHT. The AHT program consisted of 30 minute sessions, 3 days per week during 2 months. The investigators compared the effect of AHT versus no AHT, and of no AHT after 2 months versus AHT.

The endpoints were the differences in perineal tonometry, and urinary incontinence symptoms, as measured by the ICIQ_SF. Comparisons were tested with student t tests, paired or unpaired as adequate.

ELIGIBILITY:
Inclusion Criteria:

* no systematic participation in sports or physical activities (≤ 3 sessions per week, ≤ 2 weeks per month)
* between 20 and 65 years old
* with availability for three afternoons per week.

Exclusion Criteria:

* hypertension
* serious diseases
* pregnancy
* postpartum phase up to 2 months after delivery.

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-03; Primary Completion 2013-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
change of pelvic floor tone at 2 months and after 4 months | at baseline, after 2 months, and after 4 months
  Pelvic floor tone was measured by a tonometer (PhoenixTM USB2, France) in a PelvimètreTM, and results are expressed in g/cm2. A physiotherapist specialist in urogynecology did the measurement. This measure was not available for women in their first three days of menstruation or virgins

SECONDARY OUTCOMES:
change of urinary incontinence at 2 months and after 4 months | perfomed at baseline, after 2 months, and after 4 months
  Urinary incontinence was measured with the International Consultation on Incontinence Questionnaire - Short Form (ICIQ_SF) . The questionnaire includes three scored items about frequency, severity and perceived impact of incontinence.

CONTACTS AND LOCATIONS:
Overall Officials: Lidon Soriano, PhD, Principal Investigator — Alfonso X El Sabio University; Rafael J Curbelo, PhD, Principal Investigator — University of Valladolid; Loreto Carmona, PhD, Study Director — Instituto de Salud Músculo Esquelética